CLINICAL TRIAL: NCT03357835
Title: Triage With Software Assistance To Trauma Patient Who Attending To Emergency Department
Brief Title: Trauma Triage Decision With Software (TraumaDS)
Acronym: TraumaDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ahmet Akdoğan, Emergency Medicine Research Assistant, Derince Training and Research Hospital
Other Study IDs: 2017/145
Record Dates: First submitted 2017-11-13; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Trauma; Triage
Keywords: trauma; triage; software; emergency
MeSH Terms: conditions — Wounds and Injuries; Emergencies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Normal Triage: Triage scoring determined by the Ministry of Health (SB ), routinely performed by an emergency medical technician (att), will be applied when the patients are admitted to emergency services. According to this scoring, patients who need urgent care and who should not wait less than 15 minutes will be considered red coded, patients who can wait up to 60 minutes will be considered yellow coded, patients who can wait for 120 minutes or more will be considered green coded.
- Software Triage: triage maintenance / evaluation will be done with computer software called "Trauma Decision System (TraumaDS)" developed by us. As a result of the software program's direction, patients will be coded as green-yellow-orange-red area and patient care will be made in accordance with these codes. According to this scoring, patients who need urgent care and who should not wait will be considered red code, patients who should wait less than 15 minutes will be considered orange coded, patients who can wait up to 60 minutes will be considered yellow coded, patients who can wait for 120 minutes or more will be considered green coded.
  Interventions: Other: Trauma Decision System

INTERVENTIONS:
Other: Trauma Decision System — At the time of application, color codes indicating the urgency of the patients will be given according to the demographic data of the patients, the type of trauma and the vital signs were directed by the software program. As a result of the software program's direction, patients will be coded as green-yellow-orange-red area and patient care will be made in accordance with these codes.
  Groups: Software Triage

SUMMARY:
It is intended to show that a computer software called Trauma Decision System (TravmaDS) for the determination of the urgency of trauma patients who applied to Emergency Medical Clinic gives more accurate, more objective, faster results than the triage scored by medical and non-medical personnel and to show the fact that TraumaDS provides more patient satisfaction.

DETAILED DESCRIPTION:
There are limitations in our routine standard of practice in Emergency medical clinic in rapid triage about the adequacy particularly in the patient group where specific and rapid decision-making, such as trauma. The process of evaluating the patients who are directed to the green area unnecessarily in trauma care by the physician is prolonged, the evaluation process of patients who are directed to the red area unnecessarily shortens but hospital resources are being used extensively. Therefore, in this study, it was planned to perform objective triage with a computer based scoring system. Triage scoring determined by the Ministry of Health (SB ), routinely performed by an emergency medical technician (EMT), will be applied when the patients are admitted to emergency services. According to this scoring, patients who need urgent care and who should not wait less than 15 minutes will be considered red coded, patients who can wait up to 60 minutes will be considered yellow coded, patients who can wait for 120 minutes or more will be considered green coded. To the other group, triage maintenance / evaluation will be done with computer software developed by us. All patients with trauma should be included in the study, demographic data, trauma mechanism and trauma type vital signs at the time of application of the patients will be routinely observed in both groups of patients. These observations are routine for this disease group and we will not undertake any interventional procedures or screening except special routine application for research purposes. The observation and file information will be organized by the triage staff in both groups at the time of the application of the patients. In this software-based program before working on the software informative training will be given to triage staff and for this patient triage handheld computers will be given to triage staff. In order for the referring patients to be able to see the entries made with the triage software a simultaneous large-screen monitor will be used. At the time of application, color codes indicating the urgency of the patients will be given according to the demographic data of the patients, the type of trauma and the vital signs were directed by the software program. As a result of the software program's direction, patients will be coded as green-yellow-orange-red area and patient care will be made in accordance with these codes.

ELIGIBILITY:
Inclusion Criteria:

* all trauma patients who want to participate

Exclusion Criteria:

* who do not want to participate, who are not triaged, who leave the hospital before the treatment is completed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all trauma patients who want to participate in the study
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-01-31 (Estimated); Study Completion 2018-03-30 (Estimated)

PRIMARY OUTCOMES:
Difference between software triage time and traditional triage time | 5 minutes
  Investigation difference of triages made by software and normal triage

SECONDARY OUTCOMES:
30-day mortality | 30 days
  Defined as mortality within 30 days of arrival to hospital

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Akdoğan, RA, Principal Investigator — Research Assistant
Locations (1):
- Kocaeli Derince Training and Research Hospital, Derince, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided